CLINICAL TRIAL: NCT05207566
Title: Psychometric Properties of Urdu Version of Boston Carpal Tunnel Syndrome Questionnaire : A Reliability and Validity Study
Brief Title: Reliability And Validity Of Urdu Version Of Boston Carpal Tunnel Syndrome Questionnaire
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0292
Record Dates: First submitted 2022-01-24; First posted 2022-01-26 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Boston Carpal Tunnel Questionnaire; Carpal tunnel syndrome; Cultural adaptation; Validity; Urdu Version; Reliability
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Translate and culturally adapt Boston Carpal Tunnel Syndrome Questionnaire into Urdu language and find its reliability and validity in Pakistani Carpal Tunnel Syndrome patients To check its correlation with Disabilities of the Arm, Shoulder and Hand questionnaire and Visual Analog Scale.

DETAILED DESCRIPTION:
The original version of Boston Carpal Tunnel Syndrome Questionnaire will be translated into Urdu. Among idiopathic Carpal Tunnel Syndrome, 110 patients will be included in the study by convenience sampling. The selection of the patients will be done according to the criteria. Boston Carpal Tunnel Syndrome Questionnaire will be correlated with Disabilities of the Arm, Shoulder and Hand questionnaire and Visual Analog Scale and these questionnaires will be provided three times to a single patient for their assessment. Firstly, they will be provided prior to treatment and secondly just after having treatment. Thirdly, they will be given after seven days of treatment. Internal consistency and reproducibility will be used to determine reliability. Boston Carpal Tunnel Syndrome Questionnaire will be correlated with Disabilities of the Arm, Shoulder and Hand questionnaire and Visual Analog Scale to assess validity. From each patient informed consent will be obtained. Statistical Package of Social Sciences software, version 24 will be used for the analysis of data.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 18 years.
* Absence of any cognitive impairment.
* Patients having positive Tinel and Phalen test.

Exclusion Criteria:

Presence of any of following conditions.

* Diabetes
* Polyneuropathy
* Hypothyroidsm
* Rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pakistani population with CTS was included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire | 1st day
  Boston Carpal Tunnel Syndrome Questionnaireconsists of 2 subscales i.e: symptom severity & functional status.The former contains 11 items for assessing several symptoms while later contains 8 items of daily functional activities. Every item consists of 5 point score with 1 meaning no difficulty while 5 refers to severe symptoms. Boston Carpal Tunnel Syndrome Questionnaire is a short questionnaire and is completed within ten minutes
Disabilities of the Arm, Shoulder and Hand questionnaire | 1st day
  Disabilities of the Arm, Shoulder and Hand questionnaire was developed for use in problems like musculoskeletal in upper limbs. It has been translated into various languages. It consists of 30 items used to assess physical and psychosocial aspects. Every items consists of 5 point score with 1 meaning no difficulty while 5 refers to unable
Visual Analog Scale | 1st day
  VAS is used to evaluate pain and consists of a scale with 0 to 10 readings (0 meaning no pain and 10 meanings unbearable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No